CLINICAL TRIAL: NCT06988449
Title: Use of ST250 to Reconstruct Lateral Tongue Defects
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Marienhospital Stuttgart (Other)
Responsible Party: Principal Investigator, Alaa Emara, A. Professor, Cairo University
Other Study IDs: ST250 for tongue defect
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Tongue Neoplasms
Keywords: tongue defect; reconstruction; Polylactide membrane
MeSH Terms: conditions — Tongue Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tongue defect covered with ST250

SUMMARY:
To assess the use of SupraThel 250 for mucosal reconstruction in the Head & Neck region. The membrane is applied to reconstruct lateral tongue defects . healing of the mucosa and regaining of normal tongue movement and speech are assessed postoperatively.

DETAILED DESCRIPTION:
Lateral tongue defects are usually treated using radial fore-arm free grafts which require a prolonged hospital stay with higher morbidity rates. It also entails the need of multiple rehabilitation and remodeling porcdures of the transplnted flap to enable intelligible speech and tongue function.

ELIGIBILITY:
Inclusion Criteria:

* lateral tunge defects (postoncologic resection)

Exclusion Criteria:

* radio / chemotherapy
* pregnant/ breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Rickert, PhD, Principal Investigator — Marienhospital Stuttgart
Locations (1):
- MarienHospital, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarin V, Chatterjee A, Kakkar V, Juneja A. Evaluation of Tongue Functions After Free Flap Reconstruction. Indian J Otolaryngol Head Neck Surg. 2022 Oct;74(Suppl 2):2398-2403. doi: 10.1007/s12070-020-02177-1. Epub 2020 Oct 8. PMID 36452650
- See also: Related Info — https://www.thieme-connect.de/products/ejournals/conferencepdf/085434/10.1055/s-00000036.pdf